CLINICAL TRIAL: NCT03460119
Title: Use of High-Flow Nasal Cannula for Acute Respiratory Failure in the Emergency Department
Brief Title: High Flow Nasal Cannula in the Emergency Department
Acronym: HFNC
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: 3106
Record Dates: First submitted 2018-02-20; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Acute Respiratory Failure
Keywords: High Flow Nasal Cannula; Emergency department; Respiratory care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High Flow Nasal Cannula Oxygen — The high flow device that we used was an air oxygen blender (Whisper FlowⓇ), which allows FiO2 adjustment between 0.30 and 1.0 and can deliver a gas flow from 10 to 150 l/min. The gas mixture was routed from a heated humidifier (MR850 with MR 290 chamber) through a one line heated inspiratory circuit (RT241) to the subject at a temperature of 37°C via a nasal cannula (OptiflowⓇ).

SUMMARY:
The aim of this study was to describe the changes in respiratory rate, heart rate and dyspnea, before and after using HFNC in patients presenting to our emergency department with ARF.

DETAILED DESCRIPTION:
A retrospective cohort study was performed. To all adults presenting to the emergency department who used high flow nasal cannula to treat clinical signs of acute respiratory failure based on the presence of a breathing frequency ≥ 25 breath/min and increase work of breathing evidence by dyspnea, in-drawing, accessory-muscle use and/or diaphoresis despite conventional oxygen therapy ≥ 6 l/min. Demographic variables and clinical and gasometric parameters before and after two hours using HFNC were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years
* attended between July 1st, 2015 and January 31st , 2017 in the Emergency Department of the Hospital Italiano de Buenos Aires
* with clinical signs of acute respiratory failure

Exclusion Criteria:

- Pulse oximetry > 90% breathing room air

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without a history of lung disease who used high flow nasal cannula. We defined clinical signs of acute respiratory failure based on the presence of a breathing frequency ≥ 25 breath/min and increase work of breathing evidence by dyspnea, in-drawing, accessory-muscle use and/or diaphoresis, despite conventional oxygen therapy ≥ 6 l/min.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 2 hours
  The closest value of Heart Rate before starting HFNC, and two hours later was collected from the electronic clinical history.
Respiratory Rate | 2 hours
  The closest value of Respiratory Rate before starting HFNC, and two hours later was collected from the electronic clinical history.
Dyspnea | 2 hours
  The closest value of Dyspnea (Modified Borg Dyspnea scale) before starting HFNC, and two hours later was collected from the electronic clinical history. The Modified Borg Dyspnea Scale is a rated numerical score used to measure dyspnea. This scale has a minimum value of 0 ( represent no dyspnea) and a maximum value of 10 (worse dyspnea).

SECONDARY OUTCOMES:
Initial HFNC setting | 2 hours
  The gas flow rate and the fraction of inspired oxygen at the HFNC initiation of treatment were collected from the electronic clinical history.
Acute respiratory failure etiology | 3 minutes
  Presence of a breathing frequency ≥ 25 breath/min and increase work of breathing evidence by dyspnea, in-drawing, accessory-muscle use and/or diaphoresis despite conventional oxygen therapy ≥ 6 l/min.
Average time of use the HFNC | until 28 days
  The total hours of use of HFNC were collected from the electronic clinical history.
Delay of HFNC treatment | until 24hs
  The hours between the admission to HFNC initiation were collected from the electronic clinical history.
Efficacy of HFNC treatment | 28 days
  When the patient did not need for escalation to other non-invasive or invasive ventilatory support.
Failure of HFNC treatment | 28 days
  When the patient need non-invasive or invasive ventilatory support or died. The type of ventilatory support post-failure were collected from the electronic clinical history.
Mortality rate at 28 day from ED admission | 28 days
  The number of patients who died after requiring HFNCO were collected from the electronic clinical history
Palliative Care | 28 days
  Consensus between patient and/or patient´s family and the physician about the care for the terminally ill patient, provided by an organized health service

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa R Ruiz, RT, Principal Investigator — Hospital Italiano de Buenos Aires

REFERENCES:
- [Background] Roca O, Hernandez G, Diaz-Lobato S, Carratala JM, Gutierrez RM, Masclans JR; Spanish Multidisciplinary Group of High Flow Supportive Therapy in Adults (HiSpaFlow). Current evidence for the effectiveness of heated and humidified high flow nasal cannula supportive therapy in adult patients with respiratory failure. Crit Care. 2016 Apr 28;20(1):109. doi: 10.1186/s13054-016-1263-z. PMID 27121707
- [Background] El-Khatib MF. High-flow nasal cannula oxygen therapy during hypoxemic respiratory failure. Respir Care. 2012 Oct;57(10):1696-8. doi: 10.4187/respcare.02072. No abstract available. PMID 23013907
- [Background] Sztrymf B, Messika J, Mayot T, Lenglet H, Dreyfuss D, Ricard JD. Impact of high-flow nasal cannula oxygen therapy on intensive care unit patients with acute respiratory failure: a prospective observational study. J Crit Care. 2012 Jun;27(3):324.e9-13. doi: 10.1016/j.jcrc.2011.07.075. Epub 2011 Sep 29. PMID 21958974
- [Background] Ferrer M, Esquinas A, Leon M, Gonzalez G, Alarcon A, Torres A. Noninvasive ventilation in severe hypoxemic respiratory failure: a randomized clinical trial. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1438-44. doi: 10.1164/rccm.200301-072OC. Epub 2003 Sep 18. PMID 14500259
- [Background] Keenan SP, Sinuff T, Cook DJ, Hill NS. Does noninvasive positive pressure ventilation improve outcome in acute hypoxemic respiratory failure? A systematic review. Crit Care Med. 2004 Dec;32(12):2516-23. doi: 10.1097/01.ccm.0000148011.51681.e2. PMID 15599160
- [Background] Rello J, Perez M, Roca O, Poulakou G, Souto J, Laborda C, Balcells J, Serra J, Masclans JR; CRIPS investigators. High-flow nasal therapy in adults with severe acute respiratory infection: a cohort study in patients with 2009 influenza A/H1N1v. J Crit Care. 2012 Oct;27(5):434-9. doi: 10.1016/j.jcrc.2012.04.006. Epub 2012 Jul 2. PMID 22762937
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Kernick J, Magarey J. What is the evidence for the use of high flow nasal cannula oxygen in adult patients admitted to critical care units? A systematic review. Aust Crit Care. 2010 May;23(2):53-70. doi: 10.1016/j.aucc.2010.01.001. Epub 2010 Mar 5. PMID 20206546
- [Background] Messika J, Ben Ahmed K, Gaudry S, Miguel-Montanes R, Rafat C, Sztrymf B, Dreyfuss D, Ricard JD. Use of High-Flow Nasal Cannula Oxygen Therapy in Subjects With ARDS: A 1-Year Observational Study. Respir Care. 2015 Feb;60(2):162-9. doi: 10.4187/respcare.03423. Epub 2014 Nov 4. PMID 25371400
- [Background] Vargas F, Saint-Leger M, Boyer A, Bui NH, Hilbert G. Physiologic Effects of High-Flow Nasal Cannula Oxygen in Critical Care Subjects. Respir Care. 2015 Oct;60(10):1369-76. doi: 10.4187/respcare.03814. Epub 2015 May 5. PMID 25944940
- [Background] Schwabbauer N, Berg B, Blumenstock G, Haap M, Hetzel J, Riessen R. Nasal high-flow oxygen therapy in patients with hypoxic respiratory failure: effect on functional and subjective respiratory parameters compared to conventional oxygen therapy and non-invasive ventilation (NIV). BMC Anesthesiol. 2014 Aug 7;14:66. doi: 10.1186/1471-2253-14-66. eCollection 2014. PMID 25110463
- [Background] Lemiale V, Mokart D, Mayaux J, Lambert J, Rabbat A, Demoule A, Azoulay E. The effects of a 2-h trial of high-flow oxygen by nasal cannula versus Venturi mask in immunocompromised patients with hypoxemic acute respiratory failure: a multicenter randomized trial. Crit Care. 2015 Nov 2;19:380. doi: 10.1186/s13054-015-1097-0. PMID 26521922
- [Background] Sztrymf B, Messika J, Bertrand F, Hurel D, Leon R, Dreyfuss D, Ricard JD. Beneficial effects of humidified high flow nasal oxygen in critical care patients: a prospective pilot study. Intensive Care Med. 2011 Nov;37(11):1780-6. doi: 10.1007/s00134-011-2354-6. Epub 2011 Sep 27. PMID 21946925
- [Background] Lenglet H, Sztrymf B, Leroy C, Brun P, Dreyfuss D, Ricard JD. Humidified high flow nasal oxygen during respiratory failure in the emergency department: feasibility and efficacy. Respir Care. 2012 Nov;57(11):1873-8. doi: 10.4187/respcare.01575. Epub 2012 Mar 13. PMID 22417844
- [Background] Rittayamai N, Tscheikuna J, Praphruetkit N, Kijpinyochai S. Use of High-Flow Nasal Cannula for Acute Dyspnea and Hypoxemia in the Emergency Department. Respir Care. 2015 Oct;60(10):1377-82. doi: 10.4187/respcare.03837. Epub 2015 Jun 9. PMID 26060321
- [Background] Jeong JH, Kim DH, Kim SC, Kang C, Lee SH, Kang TS, Lee SB, Jung SM, Kim DS. Changes in arterial blood gases after use of high-flow nasal cannula therapy in the ED. Am J Emerg Med. 2015 Oct;33(10):1344-9. doi: 10.1016/j.ajem.2015.07.060. Epub 2015 Jul 30. PMID 26319192
- [Background] Hughes J, Doolabh A. Heated, humidified, high-flow nasal oxygen usage in the adult Emergency Department. Australas Emerg Nurs J. 2016 Nov;19(4):173-178. doi: 10.1016/j.aenj.2016.05.003. Epub 2016 Jun 6. PMID 27283891
- [Background] Jones PG, Kamona S, Doran O, Sawtell F, Wilsher M. Randomized Controlled Trial of Humidified High-Flow Nasal Oxygen for Acute Respiratory Distress in the Emergency Department: The HOT-ER Study. Respir Care. 2016 Mar;61(3):291-9. doi: 10.4187/respcare.04252. Epub 2015 Nov 17. PMID 26577199